CLINICAL TRIAL: NCT02026596
Title: Observational Study on Mechanisms and Prevention of Secondary Brain Injury in Subarachnoid Haemorrhage
Brief Title: SpareBrain - Mechanisms and Prevention of Secondary Brain Injury in Subarachnoid Haemorrhage
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TampereUH
Record Dates: First submitted 2013-11-25; First posted 2014-01-03 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: subrachnoid hemorrhage; secondary brain injury
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: * Blood samples
  * Cerebrospinal fluid samples
  * Microdialysate samples (from the extracellular fluid of the brain)
  * Tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- aSAH patients: Patients suffering from aneurysmal subarachnoid haemorrhage
  Interventions: Procedure: Magnetic resonance imaging; Procedure: Cerebral microdialysis catheter insertion

INTERVENTIONS:
Procedure: Magnetic resonance imaging
Procedure: Cerebral microdialysis catheter insertion — Is inserted only when invasive intracranial pressure monitoring is required. The same route with pressure probe is used for insertion.

SUMMARY:
Subarachnoidal hemorrhage (SAH) is a cause of long-term disability and death. Annually about 1000 people in Finland suffer from SAH, their average age being under 50 years. SAH has a mortality rate of 12 % acutely and 40 % of patients die within a month from admission to hospital. In addition, 30 % of the surviving patients remain with neurological deficits. Most survivors of the primary insult suffer from secondary injury during the first 2-3 weeks from the insult.

Despite the advances in neurosurgical and -radiological techniques and intensive care, the mortality and morbidity rates in SAH have not changed in recent years. There is still only limited understanding of the mechanisms of secondary insults causing brain injury after SAH.

In this study the investigators are aiming to clarify the timescale and mechanisms contributing to the secondary insults. The investigators also explore usability of novel biomarkers to guide treatment of the patients suffering from SAH.

DETAILED DESCRIPTION:
Subarachnoidal hemorrhage (SAH) is a cause of long-term disability and death. Annually about 1000 people in Finland suffer from SAH, their average age being under 50 years. SAH has a mortality rate of 12 % acutely and 40 % of patients die within a month from admission to hospital. In addition, 30 % of the surviving patients remain with neurological deficits. Most survivors of the primary insult suffer from secondary injury during the first 2-3 weeks from the insult.

Despite the advances in neurosurgical and -radiological techniques and intensive care, the mortality and morbidity rates in SAH have not changed in recent years. There is still only limited understanding of the mechanisms of secondary insults causing brain injury after SAH.

In this study the investigators are aiming to clarify the timescale and mechanisms contributing to the secondary insults. The investigators also explore usability of novel biomarkers to guide treatment of the patients suffering from SAH.

ELIGIBILITY:
Inclusion Criteria:

* aneurysmal subarachnoid haemorrhage

Exclusion Criteria:

* age under 18 years
* pregnant
* moribund patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from aneurysmal subarachnoid haemorrhage
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2013-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Neuroradiologically confirmed secondary injury lesions | up to 2 weeks after the primary insult
  Neuroradiological imaging (CT/MRI) is performed when clinically indicated and at 2 weeks after primary insult.

SECONDARY OUTCOMES:
Neurological outcome of the patient | 6 months
  Neurological outcome is evaluated with modified Rankin Scale at 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Länsi-Suomen Lääni, Finland